CLINICAL TRIAL: NCT03257839
Title: ARM 1: A Prospective, Multicenter, Multi-arm, Clinical Case Collection Program to Acquire Breast Image Data and Establish an Image Library of Exams for Use in Future Research Studies, Training, and Product Development Efforts.
Brief Title: Delphinus SoftVue Prospective Case Collection - ARM 1
Acronym: SV PCC ARM1
Status: Completed | Type: Observational
Sponsor: Delphinus Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DMT-2015.001 ARM 1; Protocol ID: 20151525 (Other: Western IRB)
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Breast Neoplasms
Keywords: SoftVue; Dense Breast Tissue; Breast Screening; Abnormal Breast; Normal Breast; Breast Imaging; Breast Biopsy; Mammography; Tomosynthesis; Automated Breast Ultrasound; Breast Cancer; Breast Carcinoma; Breast Tumors; Mammary Carcinoma; Malignant Breast Tumor; Mammary Neoplasm; Mammary Cancer; ABUS; AWBUS; Breast Tomography; ATUS; ABTUS; Mammogram; 3D Mammogram; 3D ABUS; 3D Breast Ultrasound; DBT; FFDM; Digital Mammography; Breast Ultrasound; Dense Breasts; Breast Density; Dense Parenchyma; Asymptomatic; Delphinus; Delphinus Medical Technologies; Screening Breast Ultrasound
MeSH Terms: conditions — Breast Neoplasms; Mammary Neoplasms, Animal | interventions — Mammography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Asymptomatic women with dense breast tissue: Healthy women presenting to enrollment sites for routine annual mammographic examinations, confirmed to have BI-RADS category c or d breast composition (density).
  Interventions: Device: Routine Full-Field Digital Mammography; Device: Routine Digital Breast Tomosynthesis; Device: Automated Whole Breast Ultrasound

INTERVENTIONS:
Device: Routine Full-Field Digital Mammography — Routine screening mammography exam, CC + MLO views.
  Other Names: FFDM, Digital Mammography, Mammography
Device: Routine Digital Breast Tomosynthesis — Routine screening tomosynthesis exam, CC + MLO views.
  Other Names: DBT, 3D Mammography, Tomosynthesis
Device: Automated Whole Breast Ultrasound — Bilateral breast ultrasound performed as an adjunct to mammography.
  Other Names: SoftVue, AWBUS, ABUS, 3D Breast Ultrasound, 3D ABUS, 3D Ultrasound, 3D US

SUMMARY:
The SoftVue™ is a whole breast ultrasound system with an automated scanning curvilinear ring-array transducer that employs UST. It is currently cleared under FDA 510(k) K123209 and K142517 for use as both a B-mode ultrasonic breast imaging system and color imaging of transmission data (sound speed and attenuation). SoftVue™ is not intended to be used as a replacement for screening mammography.

SoftVue uses non-ionizing ultrasound energy to generate tomographic image volumes of the whole breast. While the patient lays prone on a padded table with one breast comfortably submerged in a bath of warm water, a ring-shaped transducer, 22 cm in diameter, encircles the breast and pulses low-frequency sound waves through the water and into the breast tissue. More than 2000 elements in the curvilinear transducer's 360 degree array emit and receive ultrasound signals to analyze echoes from the breast anatomy in all directions, from the chest wall to the nipple. Not only does SoftVue capture data from the reflection of the sound waves off of tissue boundaries and structures within the breast, but because the transducer surrounds the whole breast, SoftVue also captures signals that are transmitted through the breast. This additional transmission data enhances the visualization of the anatomic structure of the breast tissue and is not currently available in any other commercially marketed breast ultrasound device.

This prospective, multicenter, multi-arm, clinical case collection program is IRB-approved and will be conducted in compliance with Good Clinical Practice, the Declaration of Helsinki and all applicable regulatory requirements. Arm 1 aims to collectively enroll up to 17,500 women at a total of up to 8 clinical sites. The design of this protocol is strictly limited to case collection; all investigational and statistical plans for future analyses will be prepared and registered separately, if they are applicable to the requirements of FDAAA 801.

Arm 1 is limited to the cohort of asymptomatic women, with heterogeneously or extremely dense breast parenchyma (BI-RADS breast composition category c or d). Matched triads of 2D digital mammography (FFDM), 3D digital mammography (DBT), and SoftVue automated whole breast ultrasound (SV)exams, from the same patient, with demographic information and clinical outcome data, will be collected during the same screening imaging episode. Ultrasound characteristics for all types of lesions, whether they are benign or malignant, will be collected, as well as objective and subjective breast density composition data.

The exams and clinical data accumulated in this prospective case collection (PCC) protocol will populate a database from which future investigations may be designed for peer reviewed publication, development of user training curriculums, building teaching case, and creating new marketing materials for SoftVue.A subset of exams will be sampled from Arm 1 for use in ROC Reader Study (protocol DMT-2015.002), which will be separately registered and is designed to evaluate the safety and efficacy of a new screening indication for use of SoftVue™ as an adjunct to screening mammography. The results of this ROC Reader Study will be submitted to the FDA for their consideration of a PMA application for SoftVue.

DETAILED DESCRIPTION:
MEDICAL DEVICES:

* SoftVue™ (SV) automated whole breast ultrasound system, 510(k) Cleared for B-Mode ultrasound breast imaging, manufactured by Delphinus Medical Technologies.
* SoftVue™ with device modifications (software, hardware, user-interface), safety-tested for human use to complete feasibility, verification, and validation testing as a routine part of product development and performed in accordance with FDA 21 CFR 812.2 (b), manufactured by Delphinus Medical Technologies.
* Full-field digital mammography (FFDM), FDA Approved for breast screening and diagnosis, various manufacturers.
* Digital breast tomosynthesis (DBT), FDA Approved for breast screening and diagnosis, various manufacturers.

OBJECTIVES:

* Primary: To establish a library of cases for use in future SoftVue™ research studies, user training, and marketing.
* Secondary: Determine the frequency and severity of adverse events (AEs) to further evaluate the safety of SoftVue.

ENDPOINTS:

From multiple clinical sites whichever comes first:

* Up to 17,500 total enrolled subjects
* Up to 105 total breast cancer cases detected at program entry screening
* At least 35 total discordant breast cancer cases, where FFDM is negative or benign (BI-RADS 1 or 2) but SV is incomplete (BIRADS 0) and diagnostic imaging workup of SV findings leads to breast biopsy with malignant pathology

SITES:

At least six (≥ 6) qualified clinical sites in the United States

* MQSA Certified
* Digital Breast Tomosynthesis Screening Program Implemented
* Academic, Community Hospital, or Private Practice Setting

PROJECT DESIGN AND PROCEDURES:

* Potential participants will be recruited from the group of women presenting for their annual breast imaging exams at multiple clinical sites utilizing 3D DBT and 2D FFDM (non-synthesized) for routine screening.
* Asymptomatic women with heterogeneously or extremely dense breast parenchyma (BI-RADS composition c or d), based on visual assessment of FFDM by trained site personnel, will be invited to consider volunteering to participate in the case collection program.
* All participants will complete the same routine screening FFDM + DBT evaluation for which they originally reported to the clinic, with a complete set of 2D views and 3D views.
* Eligible patients will receive SV as an adjunct to FFDM + DBT.
* A single Investigator (radiologist) at each site will perform sequential review of the same subjects FFDM, DBT, and SV images.
* FFDM will be evaluated for final parenchymal density (BI-RADS a through d) and then each exam will be assigned to one of 3 BI-RADS assessment categories (0, 1, 2) by the radiologist.
* Abnormal findings will be indicated by a BI-RADS assessment category of 0 (Incomplete)and will undergo diagnostic imaging evaluations consistent with universally accepted standards of care.
* All evaluation results, diagnosis and treatment outcomes will be recorded.
* Normal findings will be indicated by BI-RADS assessment categories of 1 or 2 (Negative or Benign) which will be associated with a management recommendation to resume routine screening in one year, unless symptoms or signs of breast cancer develop in the interim.
* All participants who are not diagnosed with breast cancer as a direct result of the program entry examinations, incidental evaluations, or interval symptoms, will return to the site in 12 months for their next annual screening exam, the results and outcome of which will be recorded.
* Cancer status for all participants will be surveyed from program entry until and including the completion of recommended follow-up.
* A case will be determined cancer negative if the participant has no findings suspicious for cancer throughout the interval between program entry and completion of annual follow-up.
* A case will be determined cancer positive if a pathological evaluation confirms a breast cancer diagnosis during the interval between program entry and completion of annual follow-up.

STATISTICAL ANALYSIS:

* Demographic characteristics (age, race, and ethnicity) and other baseline characteristics (e.g., project arm, project site, breast density, lesion-specific characteristics) will be tabulated for all participants.
* A flow diagram or table will illustrate patient disposition ("accountability of patient cohort") including reasons for ineligibility and/or unevaluability.
* Safety will be summarized for all enrolled women. With the exception of anticipated events, adverse events (AEs) and serious adverse events (SAEs), occurring from the time of enrollment (SoftVue) and for 24 hours following the conclusion of the SoftVue exam, will be recorded.
* A separate statistical plan will be developed for any future analysis that includes justification of sample size and, if applicable to the requirements of FDAAA 801, will be registered separately in order to share the results.

ELIGIBILITY:
Inclusion Criteria

* Female
* Any race or ethnicity
* Age 18 or older
* Asymptomatic
* Complete screening FFDM and DBT views
* BI-RADS density composition category c or d
* Willing to comply with protocol and follow-up recommendations as described in consent form, including the next annual screening exam in 12 months

Exclusion Criteria

* Weight exceeds 350lbs
* Currently pregnant or lactating by patient self-report
* Weeping rash, open wounds, or unhealed sores on the breast
* Bilateral mastectomy
* Unable to lay prone on the scan table for up to 15 minutes
* History of breast cancer diagnosis and/or treatment (chemotherapy, surgery, and/or radiation) in the past 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asymptomatic women with dense breast tissue
Sampling Method: Probability Sample
Enrollment: 7409 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
No Breast Cancer | 365 Days
  Non-Cancer cases, confirmed by normal or negative mammographic breast imaging (FFDM or DBT), or breast biopsy with benign pathology, after at least 365 days of follow-up
Breast Cancer | 365 Days
  Cancer cases, confirmed by breast biopsy with malignant pathology, within 365 days of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mary W Yamashita, MD, Principal Investigator — Keck School of Medicine, University of Southern California
Locations (10):
- United States (10):
  - USC Keck School of Medicine, Los Angeles, California
  - Mount Sinai Medical Center, Miami Beach, Florida
  - SouthCoast Imaging, Savannah, Georgia
  - Beaumont Dearborn Breast Care Center, Dearborn, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mercy Imaging Services, Washington, Missouri
  - Elizabeth Wende Breast Care, Rochester, New York
  - UNC Breast Imaging Center, Chapel Hill, North Carolina
  - Weinstein Imaging Associates, Pittsburgh, Pennsylvania
  - Ascension St. Elizabeth, Radiology Associates of the Fox Valley, Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tabar L, Duffy SW, Vitak B, Chen HH, Prevost TC. The natural history of breast carcinoma: what have we learned from screening? Cancer. 1999 Aug 1;86(3):449-62. PMID 10430253
- [Background] Duffy SW, Tabar L, Chen HH, Holmqvist M, Yen MF, Abdsalah S, Epstein B, Frodis E, Ljungberg E, Hedborg-Melander C, Sundbom A, Tholin M, Wiege M, Akerlund A, Wu HM, Tung TS, Chiu YH, Chiu CP, Huang CC, Smith RA, Rosen M, Stenbeck M, Holmberg L. The impact of organized mammography service screening on breast carcinoma mortality in seven Swedish counties. Cancer. 2002 Aug 1;95(3):458-69. doi: 10.1002/cncr.10765. PMID 12209737
- [Background] Duffy SW, Smith RA, Gabe R, Tabar L, Yen AM, Chen TH. Screening for breast cancer. Surg Oncol Clin N Am. 2005 Oct;14(4):671-97. doi: 10.1016/j.soc.2005.06.001. PMID 16226686
- [Background] Paci E, Duffy SW, Giorgi D, Zappa M, Crocetti E, Vezzosi V, Bianchi S, del Turco MR. Quantification of the effect of mammographic screening on fatal breast cancers: The Florence Programme 1990-96. Br J Cancer. 2002 Jul 1;87(1):65-9. doi: 10.1038/sj.bjc.6600301. PMID 12085258
- [Background] Tabar L, Duffy SW, Yen MF, Warwick J, Vitak B, Chen HH, Smith RA. All-cause mortality among breast cancer patients in a screening trial: support for breast cancer mortality as an end point. J Med Screen. 2002;9(4):159-62. doi: 10.1136/jms.9.4.159. PMID 12518005
- [Background] Swedish Organised Service Screening Evaluation Group. Effect of mammographic service screening on stage at presentation of breast cancers in Sweden. Cancer. 2007 Jun 1;109(11):2205-12. doi: 10.1002/cncr.22671. PMID 17471486
- [Background] Swedish Organised Service Screening Evaluation Group. Reduction in breast cancer mortality from organized service screening with mammography: 1. Further confirmation with extended data. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):45-51. doi: 10.1158/1055-9965.EPI-05-0349. PMID 16434585
- [Background] Swedish Organised Service Screening Evaluation Group. Reduction in breast cancer mortality from the organised service screening with mammography: 2. Validation with alternative analytic methods. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):52-6. doi: 10.1158/1055-9965.EPI-05-0953. PMID 16434586
- [Background] Hakama M, Pukkala E, Heikkila M, Kallio M. Effectiveness of the public health policy for breast cancer screening in Finland: population based cohort study. BMJ. 1997 Mar 22;314(7084):864-7. doi: 10.1136/bmj.314.7084.864. PMID 9093096
- [Background] Tabar L, Vitak B, Chen TH, Yen AM, Cohen A, Tot T, Chiu SY, Chen SL, Fann JC, Rosell J, Fohlin H, Smith RA, Duffy SW. Swedish two-county trial: impact of mammographic screening on breast cancer mortality during 3 decades. Radiology. 2011 Sep;260(3):658-63. doi: 10.1148/radiol.11110469. Epub 2011 Jun 28. PMID 21712474
- [Background] Michaelson JS, Silverstein M, Wyatt J, Weber G, Moore R, Halpern E, Kopans DB, Hughes K. Predicting the survival of patients with breast carcinoma using tumor size. Cancer. 2002 Aug 15;95(4):713-23. doi: 10.1002/cncr.10742. PMID 12209713
- [Background] Smith RA, Duffy SW, Gabe R, Tabar L, Yen AM, Chen TH. The randomized trials of breast cancer screening: what have we learned? Radiol Clin North Am. 2004 Sep;42(5):793-806, v. doi: 10.1016/j.rcl.2004.06.014. PMID 15337416
- [Background] Kolb TM, Lichy J, Newhouse JH. Comparison of the performance of screening mammography, physical examination, and breast US and evaluation of factors that influence them: an analysis of 27,825 patient evaluations. Radiology. 2002 Oct;225(1):165-75. doi: 10.1148/radiol.2251011667. PMID 12355001
- [Background] Kerlikowske K, Grady D, Barclay J, Sickles EA, Ernster V. Effect of age, breast density, and family history on the sensitivity of first screening mammography. JAMA. 1996 Jul 3;276(1):33-8. PMID 8667536
- [Background] Pisano ED, Gatsonis C, Hendrick E, Yaffe M, Baum JK, Acharyya S, Conant EF, Fajardo LL, Bassett L, D'Orsi C, Jong R, Rebner M; Digital Mammographic Imaging Screening Trial (DMIST) Investigators Group. Diagnostic performance of digital versus film mammography for breast-cancer screening. N Engl J Med. 2005 Oct 27;353(17):1773-83. doi: 10.1056/NEJMoa052911. Epub 2005 Sep 16. PMID 16169887
- [Background] Cole EB, Pisano ED, Kistner EO, Muller KE, Brown ME, Feig SA, Jong RA, Maidment AD, Staiger MJ, Kuzmiak CM, Freimanis RI, Lesko N, Rosen EL, Walsh R, Williford M, Braeuning MP. Diagnostic accuracy of digital mammography in patients with dense breasts who underwent problem-solving mammography: effects of image processing and lesion type. Radiology. 2003 Jan;226(1):153-60. doi: 10.1148/radiol.2261012024. PMID 12511684
- [Background] Haas BM, Kalra V, Geisel J, Raghu M, Durand M, Philpotts LE. Comparison of tomosynthesis plus digital mammography and digital mammography alone for breast cancer screening. Radiology. 2013 Dec;269(3):694-700. doi: 10.1148/radiol.13130307. Epub 2013 Oct 28. PMID 23901124
- [Background] Svahn TM, Chakraborty DP, Ikeda D, Zackrisson S, Do Y, Mattsson S, Andersson I. Breast tomosynthesis and digital mammography: a comparison of diagnostic accuracy. Br J Radiol. 2012 Nov;85(1019):e1074-82. doi: 10.1259/bjr/53282892. Epub 2012 Jun 6. PMID 22674710
- [Background] Rafferty EA, Park JM, Philpotts LE, Poplack SP, Sumkin JH, Halpern EF, Niklason LT. Assessing radiologist performance using combined digital mammography and breast tomosynthesis compared with digital mammography alone: results of a multicenter, multireader trial. Radiology. 2013 Jan;266(1):104-13. doi: 10.1148/radiol.12120674. Epub 2012 Nov 20. PMID 23169790
- [Background] Wolfe JN. Breast patterns as an index of risk for developing breast cancer. AJR Am J Roentgenol. 1976 Jun;126(6):1130-7. doi: 10.2214/ajr.126.6.1130. PMID 179369
- [Background] Ursin G, Hovanessian-Larsen L, Parisky YR, Pike MC, Wu AH. Greatly increased occurrence of breast cancers in areas of mammographically dense tissue. Breast Cancer Res. 2005;7(5):R605-8. doi: 10.1186/bcr1260. Epub 2005 Jun 8. PMID 16168104
- [Background] Titus-Ernstoff L, Tosteson AN, Kasales C, Weiss J, Goodrich M, Hatch EE, Carney PA. Breast cancer risk factors in relation to breast density (United States). Cancer Causes Control. 2006 Dec;17(10):1281-90. doi: 10.1007/s10552-006-0071-1. PMID 17111260
- [Background] Boyd NF, Guo H, Martin LJ, Sun L, Stone J, Fishell E, Jong RA, Hislop G, Chiarelli A, Minkin S, Yaffe MJ. Mammographic density and the risk and detection of breast cancer. N Engl J Med. 2007 Jan 18;356(3):227-36. doi: 10.1056/NEJMoa062790. PMID 17229950
- [Background] Boyd NF, Martin LJ, Yaffe MJ, Minkin S. Mammographic density: a hormonally responsive risk factor for breast cancer. J Br Menopause Soc. 2006 Dec;12(4):186-93. doi: 10.1258/136218006779160436. PMID 17178021
- [Background] Torres-Mejia G, De Stavola B, Allen DS, Perez-Gavilan JJ, Ferreira JM, Fentiman IS, Dos Santos Silva I. Mammographic features and subsequent risk of breast cancer: a comparison of qualitative and quantitative evaluations in the Guernsey prospective studies. Cancer Epidemiol Biomarkers Prev. 2005 May;14(5):1052-9. doi: 10.1158/1055-9965.EPI-04-0717. PMID 15894652
- [Background] Stone J, Dite GS, Gunasekara A, English DR, McCredie MR, Giles GG, Cawson JN, Hegele RA, Chiarelli AM, Yaffe MJ, Boyd NF, Hopper JL. The heritability of mammographically dense and nondense breast tissue. Cancer Epidemiol Biomarkers Prev. 2006 Apr;15(4):612-7. doi: 10.1158/1055-9965.EPI-05-0127. PMID 16614099
- [Background] Kolb TM, Lichy J, Newhouse JH. Occult cancer in women with dense breasts: detection with screening US--diagnostic yield and tumor characteristics. Radiology. 1998 Apr;207(1):191-9. doi: 10.1148/radiology.207.1.9530316.
- [Background] Checka CM, Chun JE, Schnabel FR, Lee J, Toth H. The relationship of mammographic density and age: implications for breast cancer screening. AJR Am J Roentgenol. 2012 Mar;198(3):W292-5. doi: 10.2214/AJR.10.6049. PMID 22358028
- [Background] Sprague BL, Gangnon RE, Burt V, Trentham-Dietz A, Hampton JM, Wellman RD, Kerlikowske K, Miglioretti DL. Prevalence of mammographically dense breasts in the United States. J Natl Cancer Inst. 2014 Sep 12;106(10):dju255. doi: 10.1093/jnci/dju255. Print 2014 Oct. PMID 25217577
- [Background] Rieber A, Brambs HJ, Gabelmann A, Heilmann V, Kreienberg R, Kuhn T. Breast MRI for monitoring response of primary breast cancer to neo-adjuvant chemotherapy. Eur Radiol. 2002 Jul;12(7):1711-9. doi: 10.1007/s00330-001-1233-x. Epub 2002 Feb 14. PMID 12111062
- [Background] King V, Brooks JD, Bernstein JL, Reiner AS, Pike MC, Morris EA. Background parenchymal enhancement at breast MR imaging and breast cancer risk. Radiology. 2011 Jul;260(1):50-60. doi: 10.1148/radiol.11102156. Epub 2011 Apr 14. PMID 21493794
- [Background] Saslow D, Boetes C, Burke W, Harms S, Leach MO, Lehman CD, Morris E, Pisano E, Schnall M, Sener S, Smith RA, Warner E, Yaffe M, Andrews KS, Russell CA; American Cancer Society Breast Cancer Advisory Group. American Cancer Society guidelines for breast screening with MRI as an adjunct to mammography. CA Cancer J Clin. 2007 Mar-Apr;57(2):75-89. doi: 10.3322/canjclin.57.2.75. PMID 17392385
- [Background] Kuhl CK, Schrading S, Strobel K, Schild HH, Hilgers RD, Bieling HB. Abbreviated breast magnetic resonance imaging (MRI): first postcontrast subtracted images and maximum-intensity projection-a novel approach to breast cancer screening with MRI. J Clin Oncol. 2014 Aug 1;32(22):2304-10. doi: 10.1200/JCO.2013.52.5386. Epub 2014 Jun 23. PMID 24958821
- [Background] Corsetti V, Ferrari A, Ghirardi M, Bergonzini R, Bellarosa S, Angelini O, Bani C, Ciatto S. Role of ultrasonography in detecting mammographically occult breast carcinoma in women with dense breasts. Radiol Med. 2006 Apr;111(3):440-8. doi: 10.1007/s11547-006-0040-5. Epub 2006 Apr 11. English, Italian. PMID 16683089
- [Background] Crystal P, Strano SD, Shcharynski S, Koretz MJ. Using sonography to screen women with mammographically dense breasts. AJR Am J Roentgenol. 2003 Jul;181(1):177-82. doi: 10.2214/ajr.181.1.1810177. PMID 12818853
- [Background] Berg WA, Zhang Z, Lehrer D, Jong RA, Pisano ED, Barr RG, Bohm-Velez M, Mahoney MC, Evans WP 3rd, Larsen LH, Morton MJ, Mendelson EB, Farria DM, Cormack JB, Marques HS, Adams A, Yeh NM, Gabrielli G; ACRIN 6666 Investigators. Detection of breast cancer with addition of annual screening ultrasound or a single screening MRI to mammography in women with elevated breast cancer risk. JAMA. 2012 Apr 4;307(13):1394-404. doi: 10.1001/jama.2012.388. PMID 22474203
- [Background] Hooley RJ, Greenberg KL, Stackhouse RM, Geisel JL, Butler RS, Philpotts LE. Screening US in patients with mammographically dense breasts: initial experience with Connecticut Public Act 09-41. Radiology. 2012 Oct;265(1):59-69. doi: 10.1148/radiol.12120621. Epub 2012 Jun 21. PMID 22723501
- [Background] Kelly KM, Dean J, Comulada WS, Lee SJ. Breast cancer detection using automated whole breast ultrasound and mammography in radiographically dense breasts. Eur Radiol. 2010 Mar;20(3):734-42. doi: 10.1007/s00330-009-1588-y. Epub 2009 Sep 2. PMID 19727744
- [Background] Corsetti V, Houssami N, Ferrari A, Ghirardi M, Bellarosa S, Angelini O, Bani C, Sardo P, Remida G, Galligioni E, Ciatto S. Breast screening with ultrasound in women with mammography-negative dense breasts: evidence on incremental cancer detection and false positives, and associated cost. Eur J Cancer. 2008 Mar;44(4):539-44. doi: 10.1016/j.ejca.2008.01.009. Epub 2008 Feb 11. PMID 18267357
- [Background] Leconte I, Feger C, Galant C, Berliere M, Berg BV, D'Hoore W, Maldague B. Mammography and subsequent whole-breast sonography of nonpalpable breast cancers: the importance of radiologic breast density. AJR Am J Roentgenol. 2003 Jun;180(6):1675-9. doi: 10.2214/ajr.180.6.1801675. PMID 12760942
- [Background] Kaplan SS. Clinical utility of bilateral whole-breast US in the evaluation of women with dense breast tissue. Radiology. 2001 Dec;221(3):641-9. doi: 10.1148/radiol.2213010364. PMID 11719658
- [Background] Buchberger W, Niehoff A, Obrist P, DeKoekkoek-Doll P, Dunser M. Clinically and mammographically occult breast lesions: detection and classification with high-resolution sonography. Semin Ultrasound CT MR. 2000 Aug;21(4):325-36. doi: 10.1016/s0887-2171(00)90027-1. PMID 11014255
- [Background] Gordon PB, Goldenberg SL. Malignant breast masses detected only by ultrasound. A retrospective review. Cancer. 1995 Aug 15;76(4):626-30. doi: 10.1002/1097-0142(19950815)76:43.0.co;2-z. PMID 8625156
- [Background] Berg WA, Blume JD, Cormack JB, Mendelson EB, Lehrer D, Bohm-Velez M, Pisano ED, Jong RA, Evans WP, Morton MJ, Mahoney MC, Larsen LH, Barr RG, Farria DM, Marques HS, Boparai K; ACRIN 6666 Investigators. Combined screening with ultrasound and mammography vs mammography alone in women at elevated risk of breast cancer. JAMA. 2008 May 14;299(18):2151-63. doi: 10.1001/jama.299.18.2151. PMID 18477782
- [Background] Berg WA, Blume JD, Cormack JB, Mendelson EB. Operator dependence of physician-performed whole-breast US: lesion detection and characterization. Radiology. 2006 Nov;241(2):355-65. doi: 10.1148/radiol.2412051710. PMID 17057064
- [Background] Brem RF, Tabar L, Duffy SW, Inciardi MF, Guingrich JA, Hashimoto BE, Lander MR, Lapidus RL, Peterson MK, Rapelyea JA, Roux S, Schilling KJ, Shah BA, Torrente J, Wynn RT, Miller DP. Assessing improvement in detection of breast cancer with three-dimensional automated breast US in women with dense breast tissue: the SomoInsight Study. Radiology. 2015 Mar;274(3):663-73. doi: 10.1148/radiol.14132832. Epub 2014 Oct 17. PMID 25329763
- [Background] Ranger B, Littrup PJ, Duric N, Chandiwala-Mody P, Li C, Schmidt S, Lupinacci J. Breast ultrasound tomography versus MRI for clinical display of anatomy and tumor rendering: preliminary results. AJR Am J Roentgenol. 2012 Jan;198(1):233-9. doi: 10.2214/AJR.11.6910. PMID 22194502
- [Background] Mandelson MT, Oestreicher N, Porter PL, White D, Finder CA, Taplin SH, White E. Breast density as a predictor of mammographic detection: comparison of interval- and screen-detected cancers. J Natl Cancer Inst. 2000 Jul 5;92(13):1081-7. doi: 10.1093/jnci/92.13.1081. PMID 10880551
- [Background] Houssami N, Irwig L, Ciatto S. Radiological surveillance of interval breast cancers in screening programmes. Lancet Oncol. 2006 Mar;7(3):259-65. doi: 10.1016/S1470-2045(06)70617-9. PMID 16510335
- [Background] Roubidoux MA, Bailey JE, Wray LA, Helvie MA. Invasive cancers detected after breast cancer screening yielded a negative result: relationship of mammographic density to tumor prognostic factors. Radiology. 2004 Jan;230(1):42-8. doi: 10.1148/radiol.2301020589. PMID 14695385
- See also: Delphinus Medical Technologies — https://www.delphinusmt.com/